CLINICAL TRIAL: NCT06183346
Title: Global Evaluation of Cholecystectomy Knowledge and Outcomes
Brief Title: Global Evaluation of Cholecystectomy Knowledge and Outcomes, Indonesia
Acronym: GECKO-ID
Status: Completed | Type: Observational
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Christopher Ryalino, MD, Principal Investigator, Udayana University
Other Study IDs: GECKO-INDONESIA
Record Dates: First submitted 2023-07-14; First posted 2023-12-27 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Cholecystectomy
Keywords: surgery; cholecystectomy; robotic; audit; international; multicentre; prospective; observational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Main Cohort (Single Cohort): The main cohort consists of all patients who will undergo either emergency/urgent/delayed/elective cholecystectomy in all participating hospitals in Indonesia. Inclusion/exclusion criteria will be applied.

SUMMARY:
GECKO is a prospective, international, multicentre, observational cohort study delivered by GlobalSurg Collaborative. This will be on consecutive patients undergoing cholecystectomy, between 31st July 2023 to 19th November 2023, with follow-up at 30-day and one-year postoperatively. Mini-teams of up to five collaborators per 14-day data collection period will prospectively collect data at each participating centre.

The primary aim is to define the global variation in compliance to pre-, intra-, and post-operative audit standards. The subjects will be observed and interviewed during pre-surgery hospitalization up to one-year post-surgery.

DETAILED DESCRIPTION:
Audit Standards include:

1. Pre-operative

   * Interventional radiology service
   * Risk Stratification (Tokyo Guidelines).
   * Timing of surgery
2. Intraoperative

   * Critical Safety View (CVS)
   * Intraoperative imaging
   * Bailout Procedures
   * Antibiotic use
   * Use of drains
   * Bile Duct Injury (BDI)
3. Postoperative

   * 30-day readmission
   * Critical Care

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (greater than or including 18 years of age)
* Undergo primary cholecystectomy (as the main procedure)
* Any open, laparoscopic, robotic approaches are eligible
* Elective, delayed and emergency cholecystectomy

Exclusion Criteria:

* Cholecystectomy as a part of another surgical procedure (Whipple's, bariatric, transplant)
* Patients with Mirizzi syndrome
* Patients returning to theatre and requiring a cholecystectomy for whatever indication
* Known gallbladder malignancy: Gallbladder cancer diagnosed preoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing cholecystectomy, between 31st July - 19th November 2023, with follow-up at 30-day and one-year postoperatively
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days after the surgery
  All-cause mortality rate at 30-days after cholecystectomy, assessed as dichotomous variable (survivor vs non-survivor)
1-year mortality | 1 year after the surgery
  All-cause mortality rate at 1-year after cholecystectomy, assessed as dichotomous variable (survivor vs non-survivor)

SECONDARY OUTCOMES:
Critical care admission | 24 hours after the surgery
  All-cause ICU admission rate at 24-hours after cholecystectomy, assessed as dichotomous variable (yes vs no)
30-day readmission | 30 days after surgery
  All-cause readmission rate at 30-days after cholecystectomy, assessed as dichotomous variable (yes vs no)

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - RSUP Prof. Ngoerah, Denpasar, Bali
  - RS Universitas Udayana, Jimbaran, Bali

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website for International GECKO study — https://www.globalsurgeryunit.org/clinical-trials-holding-page/project-gecko/